CLINICAL TRIAL: NCT01524289
Title: A 1-Year, Worldwide, Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled Study to Assess the Efficacy and Tolerability of Anacetrapib When Added to Ongoing Statin Therapy With or Without Other Lipid Modifying Medication(s) in Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: Study to Assess the Tolerability and Efficacy of Anacetrapib (MK-0859) Co-Administered With Statin in Participants With Heterozygous Familial Hypercholesterolemia (MK-0859-020)
Acronym: REALIZE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-020; 2011-004525-27 (EudraCT Number); MK-0859-020 (Other: Merck)
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Hyperlipoproteinemia Type II; Hypercholesterolemia, Familial
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anacetrapib (Experimental): Participants were administered one tablet of 100 mg anacetrapib orally once daily with a meal for 52 weeks during the treatment period.
  Interventions: Drug: Anacetrapib
- Placebo (Placebo Comparator): Participants were administered one matching placebo tablet orally once daily with a meal for 52 weeks during the treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anacetrapib — One oral tablet, orally once daily for 52 weeks
  Other Names: MK-0859
  Arms: Anacetrapib
Drug: Placebo — One oral tablet once daily for 52 weeks
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and tolerability of adding anacetrapib to ongoing statin therapy in participants with heterozygous familial hypercholesterolemia (HeFH).

ELIGIBILITY:
Inclusion Criteria:

* If of reproductive potential, must agree to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control for the duration of the study
* Diagnosed with Heterozygous Familial Hypercholesterolemia (HeFH)
* Have been treated with an optimal dose of statin for at least 6 weeks

Exclusion Criteria:

* Received treatment with low-density lipoprotein (LDL) apheresis within 4 weeks of screening or expect to undergo treatment with LDL apheresis during the course of the study
* Homozygous familial hypercholesterolemia
* Severe chronic heart failure
* Uncontrolled hypertension
* Uncontrolled cardiac arrhythmias, myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG), unstable angina, or stroke within 3 months
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Active or chronic hepatobiliary, hepatic, or gall bladder disease
* Pregnant or breast-feeding, or plans to become pregnant during the study or within 2 years after stopping study medication
* History of ileal bypass, gastric bypass, or other significant condition associated with malabsorption
* Human immunodeficiency virus (HIV) positive
* History of malignancy ≤5 years
* Donated blood products or has had phlebotomy of >300 mL within 8 weeks or intends to donate 250 mL of blood products or receive blood products within the projected duration of the study
* Currently taking medications that are potent inhibitors or inducers of cytochrome P450 3A4 (CYP3A) (including but not limited to cyclosporine, systemic itraconazole or ketoconazole, erythromycin, clarithromycin, or telithromycin, nefazodone, protease inhibitors, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St John's wort) or has discontinued treatment <3 weeks prior
* Consumes more than 2 alcoholic drinks per day
* Currently participating or has participated in a study with an investigational compound or device within 3 months
* Receiving treatment with systemic corticosteroids or taking systemic anabolic agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2012-02-03 (Actual); Primary Completion 2014-02-12 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Kastelein JJ, Besseling J, Shah S, Bergeron J, Langslet G, Hovingh GK, Al-Saady N, Koeijvoets M, Hunter J, Johnson-Levonas AO, Fable J, Sapre A, Mitchel Y. Anacetrapib as lipid-modifying therapy in patients with heterozygous familial hypercholesterolaemia (REALIZE): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet. 2015 May 30;385(9983):2153-61. doi: 10.1016/S0140-6736(14)62115-2. Epub 2015 Mar 3. PMID 25743173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 26 study centers. Participants were to complete a 2-week placebo run-in period, a 52-week randomized treatment phase and a 12-week reversal phase (safety follow-up).
Pre-assignment Details: The study enrolled participants who were 18 to 80 years old, had a genotype-confirmed or clinical diagnosis of heterozygous familial hypercholesterolemia (HeFH), and had been treated with an optimal dose of statin for at least 6 weeks.
Groups:
- Anacetrapib 100 mg: Participants were administered one tablet of 100 mg anacetrapib orally once daily with a meal for 52 weeks during the treatment phase.
- Placebo: Participants were administered one matching placebo tablet orally once daily with a meal for 52 weeks during the treatment phase.
Period: Overall Study
Arm/Group | Anacetrapib 100 mg | Placebo
Started | 204 | 102
Treated | 203 | 102
Completed | 174 | 88
Not Completed | 30 | 14
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 5 | 1
Not completed — Withdrawal by Subject | 11 | 7
Not completed — Adverse Event | 12 | 5
Not completed — Did not take study medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anacetrapib 100 mg | Placebo | Total
Number analyzed (Participants) | 204 | 102 | 306
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (11.8) | 55.7 (11.9) | 55.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 52 | 136
  Male | 120 | 50 | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black or African American | 0 | 1 | 1
  Multi-racial | 3 | 1 | 4
  White | 199 | 100 | 299

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) - Treatment Phase
Description: LDL-C levels were measured at baseline and week 52 (or at discontinuation) using a beta quantification method. The Treatment Phase was the period from the date of the participant's first dose of study treatment (randomization visit, Visit 3) to the participant's last visit on treatment (discontinuation visit or Visit 8 [Week 52]).
Time Frame: Baseline and Week 52
Population: The full analysis set (FAS) population consisted of all randomized participants who received at least one dose of study treatment, had at least one post randomization observation for the analysis endpoint subsequent to at least one dose of study treatment and had baseline data for those analyses that require baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 165 | 85
Percent Change | -36.0 [-39.5 to -32.5] | 3.7 [-1.2 to 8.6]
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Between group comparison of percent change from baseline performed using Constrained Longitudinal Data Analysis (cLDA) model; Difference in Least Squares (LS) Means = -39.7, 95% CI 2-sided [-45.7 to -33.7]

2. Primary Outcome: Percentage of Participants With Any Adverse Event - Treatment Phase
Description: An adverse event (AE) or experience was any unfavorable and unintended change in the structure (signs), function (symptoms), or chemistry (laboratory data) of the body temporally associated with any use of a study treatment, whether or not considered related to the use of the study treatment. Any worsening of a preexisting condition which was temporally associated with the use of the study treatment is also an AE. The percentage of participants with any adverse event during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: The all participants as treated (APaT) population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 203 | 102
Percentage of Participants | 76.4 | 78.4
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; Difference in Percentages = -2.1, 95% CI 2-sided [-11.5 to 8.4]; Miettinen and Nurminen

3. Primary Outcome: Percentage of Participants With Any Treatment-Related Adverse Event - Treatment Phase
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of the treatment. Any worsening of a preexisting condition which was temporally associated with the use of the study treatment was also an AE. AEs reported by the investigator as definitely, probably or possibly related to study treatment were considered treatment-related. The percentage of participants with any treatment-related adverse event during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: The APaT population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 203 | 102
Percentage of Participants | 18.2 | 13.7
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; Difference in Percentages = 4.5, 95% CI 2-sided [-4.8 to 12.6]; Miettinen and Nurminen

4. Primary Outcome: Percentage of Participants With Any Serious Adverse Event - Treatment Phase
Description: A serious adverse experience (SAE) was any adverse event that occurred at any dose that resulted in death or was life threatening, resulted in a persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, or was a congenital anomaly/birth defect. The percentage of participants with any serious adverse event during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: The APaT population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 203 | 102
Percentage of Participants | 8.9 | 9.8
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; Difference in Percentages = -0.9, 95% CI 2-sided [-8.9 to 5.6]; Miettinen & Nurminen

5. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an Adverse Event - Treatment Phase
Description: An adverse event (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of the drug. Any worsening of a preexisting condition which was temporally associated with the use of the study drug was also an AE. The percentage of participants who discontinued study treatment due to an AE during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: The APaT population consists of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 203 | 102
Percentage of Participants | 5.9 | 4.9
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; Difference in Percentages = 1.0, 95% CI 2-sided [-5.5 to 6.1]; Miettinen and Nurminen

6. Primary Outcome: Percentage of Participants With Changes in Systolic Blood Pressure (SBP) >= 10 mm Hg
Description: Participants had SBP assessed at baseline and throughout the 52-week treatment period. Percentage of participants who had a SBP reading that was >= 10 mm Hg higher than their baseline SBP for any assessment performed during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment and had at least one post-baseline test result that met pre-determined criteria.
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 45.0 | 53.5
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-Specified; p = 0.168, Miettinen and Nurminen; Difference in Percentages = -8.4, 95% CI 2-sided [-20.1 to 3.5]

7. Primary Outcome: Percentage of Participants With Changes in SBP >= 15 mm Hg
Description: Participants had SBP assessed at baseline and throughout the 52-week treatment period. The percentage of participants who had a SBP reading that was >= 15 mm Hg higher than their baseline SBP for any assessment performed during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 26.2 | 33.7
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.179, Miettinen and Nurminen; Difference in Percentages = -7.4, 95% CI 2-sided [-18.7 to 3.3]

8. Primary Outcome: Percentage of Participants With Changes in Diastolic Blood Pressure (DBP) >= 10 mm Hg
Description: Participants had DBP assessed at baseline and throughout the 52-week treatment period. The percentage of participants who had a DBP reading that was >= 10 mm Hg higher than their baseline DBP for any assessment performed during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 22.8 | 36.6
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.011, Miettinen and Nurminen; Difference in Percentages = -13.9, 95% CI 2-sided [-25.0 to -3.1]

9. Primary Outcome: Percentage of Participants With Sodium Levels > Upper Limit of Normal (ULN)
Description: Participants had sodium levels assessed throughout the 52-week treatment period. The percentage of participants who had any sodium level that was greater than the ULN of 145 mEq/L during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 11.4 | 9.9
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.696, Miettinen and Nurminen; Difference in Percentages = 1.5, 95% CI 2-sided [-6.8 to 8.4]

10. Primary Outcome: Percentage of Participants With Chloride Levels > ULN
Description: Participants had chloride levels assessed throughout the 52-week treatment period. The percentage of participants who had any chloride level that was > the ULN of 110 mEq/L during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 0.5 | 0.0
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.480, Miettinen and Nurminen; Difference in Percentages = 0.5, 95% CI 2-sided [-3.2 to 2.8]

11. Primary Outcome: Percentage of Participants With Potassium Levels < Lower Limit of Normal (LLN)
Description: Participants had potassium levels assessed throughout the 52-week treatment period. The percentage of participants who had any potassium level that was < the LLN of 3.5 mEq/L during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 1.5 | 1.0
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.722, Miettinen and Nurminen; Difference in Percentages = 0.5, 95% CI 2-sided [-4.0 to 3.5]

12. Primary Outcome: Percentage of Participants With Bicarbonate Levels > ULN
Description: Participants had bicarbonate levels assessed throughout the 52-week treatment period. The percentage of participants who had any bicarbonate level that was > the ULN of 33 mEq/L during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p > 0.999, Miettinen and Nurminen; Difference in Percentages = 0.0, 95% CI 2-sided [-3.7 to 1.9]

13. Primary Outcome: Percentage of Participants With Consecutive Changes in Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) of >=3 x ULN
Description: Participants had AST and ALT levels assessed throughout the 52-week treatment period. The percentage of participants who had 2 consecutive assessments of either AST or ALT that were 3 x ULN or greater during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 1.5 | 1.0
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.722, Miettinen and Nurminen; Difference in Percentages = 0.5, 95% CI 2-sided [-4.0 to 3.5]

14. Primary Outcome: Percentage of Participants With Creatine Kinase (CK) Level >=10 x ULN
Description: Participants had CK levels assessed throughout the 52-week treatment period. The percentage of participants who had any CK level that was >=10 x ULN during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 0.0 | 1.0
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.157, Miettinen and Nurminen; Difference in Percentages = -1.0, 95% CI 2-sided [-5.4 to 0.9]

15. Primary Outcome: Percentage of Participants With CK Level >=10 x ULN With Muscle Spasms
Description: Participants had CK levels assessed throughout the 52-week treatment period. The percentage of participants who had any CK level that was >=10 x ULN and had associated muscle spasms during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 202 | 101
Percentage of Participants | 0.0 | 1.0
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.157, Miettinen and Nurminen; Difference in Percentages = -1.0, 95% CI 2-sided [-5.4 to 0.9]

16. Primary Outcome: Percentage of Participants Adjudicated Cardiovascular (CV) SAE
Description: An AE or suspected adverse reaction was considered an SAE if it resulted in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. All events were adjudicated by an expert committee independent of the Sponsor. The percentage of participants that experienced adjudicated SAEs of CV death, non-fatal stroke, non-fatal myocardial infarction, or unstable angina during the treatment phase is presented.
Time Frame: Up to 52 weeks
Population: The APaT population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 203 | 102
Percentage of Participants | 1.5 | 0.0
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p = 0.218, Miettinen and Nurminen; Difference in Percentages = 1.5, 95% CI 2-sided [-2.2 to 4.3]

17. Primary Outcome: Percentage of Participants Who Died From Any Cause - Treatment Phase
Description: The percentage of participants who died from any cause during the treatment phase is presented. All deaths were adjudicated by an expert committee independent of the Sponsor.
Time Frame: Up to 52 weeks
Population: The APaT population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 203 | 102
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Other — Pre-specified; p > 0.999, Miettinen and Nurminen; Difference in Percentages = 0.0, 95% CI 2-sided [-3.6 to 1.9]

18. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol Levels
Description: The efficacy of adding anacetrapib 100 mg relative to placebo on plasma concentrations of high-density lipoprotein cholesterol (HDL-C) was evaluated at Week 0 (start of treatment phase) and Week 52 (end of treatment phase) or at discontinuation.
Time Frame: Baseline and Week 52
Population: The FAS population consisted of all randomized participants who received at least one dose of study treatment and had at least one post randomization observation for the analysis endpoint subsequent to at least one dose of study treatment, and had baseline data for those analyses that require baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 173 | 88
Percent Change | 105.8 [101.1 to 110.6] | 3.7 [-2.8 to 10.3]
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares (LS) Means = 102.1, 95% CI 2-sided [94.2 to 110.1]

19. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol Levels
Description: The efficacy of adding anacetrapib 100 mg was evaluated relative to placebo on plasma concentrations of non-high-density lipoprotein cholesterol (HDL-C) for the FAS population at Week 0 (start of treatment phase) and Week 52 (end of treatment phase) or at discontinuation.
Time Frame: Baseline and Week 52
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 173 | 88
Percent Change | -32.0 [-35.1 to -28.9] | 4.4 [0.1 to 8.8]
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in LS Means = -36.4, 95% CI 2-sided [-41.7 to -31.1]

20. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B Levels
Description: The efficacy of adding anacetrapib 100 mg was evaluated relative to placebo on plasma concentrations of apolipoprotein (Apo) B for the FAS population at Week 0 (start of treatment phase) and Week 52 (end of treatment phase) or at discontinuation.
Time Frame: Baseline and Week 52
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Percent Change
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 173 | 88
Percent Change | -19.6 [-22.5 to -16.8] | 5.2 [1.3 to 9.1]
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in LS Means = -24.8, 95% CI 2-sided [-29.5 to -20.1]

21. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) A-1 Levels
Description: The efficacy of adding anacetrapib 100 mg was evaluated relative to placebo on plasma concentrations of Apo A-1 for the FAS population at Week 0 (start of treatment phase) and Week 52 (end of treatment phase) or at discontinuation.
Time Frame: Baseline and Week 52
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Percent Change
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 173 | 88
Percent Change | 35.8 [33.0 to 38.6] | 2.9 [-1.0 to 6.8]
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in LS Means = 32.9, 95% CI 2-sided [28.2 to 37.6]

22. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) (Lp[a]) Levels
Description: The efficacy of adding anacetrapib 100 mg was evaluated relative to placebo on plasma concentrations of lipoprotein(a) (Lp[a]) for the FAS population at Week 0 (start of treatment phase) and Week 52 (end of treatment phase) or at discontinuation.
Time Frame: Baseline and Week 52
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Percent Change
Arm/Group | Anacetrapib 100 mg | Placebo
Number analyzed (Participants) | 174 | 88
Percent Change | -31.8 [-37.4 to -26.3] | 0.0 [-5.1 to 5.1]
Statistical Analysis 1: Comparison: Anacetrapib 100 mg vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -27.9, 95% CI 2-sided [-34.7 to -21.2] — Hodges-Lehmann estimate of the median difference between treatments with a corresponding distribution-free confidence interval (CI) based on Wilcoxon's rank sum test

ADVERSE EVENTS:
Time Frame: Up to 64 weeks
Description: Safety population: All participants who received at least 1 dose of study treatment. The treatment phase included AEs reported during the 52-week period from the date of the first dose of study treatment to the last visit on treatment (discontinuation visit or Week 52). The reversal phase included AEs reported during the 12-week period from the day after the treatment phase to the last visit (discontinuation or Week 64).
Groups:
- Anacetrapib 100 mg - Treatment Phase: Participants were administered one tablet of 100 mg anacetrapib orally once daily with a meal for 52 weeks.
- Placebo - Treatment Phase: Participants were administered one matching placebo tablet orally once daily with a meal for 52 weeks.
- Anacetrapib 100 mg - Reversal Phase; Placebo - Reversal Phase: Safety data that was reported during the 12-week period from the day after the treatment phase to the participant's last visit (discontinuation visit or week 64).
Arm/Group | Anacetrapib 100 mg - Treatment Phase | Placebo - Treatment Phase | Anacetrapib 100 mg - Reversal Phase | Placebo - Reversal Phase
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/102 | 0/196 | 0/95
Serious Adverse Events (participants affected / at risk) | 18/203 | 10/102 | 3/196 | 2/95
Other Adverse Events (participants affected / at risk) | 87/203 | 41/102 | 0/196 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anacetrapib 100 mg - Treatment Phase (N=203) | Placebo - Treatment Phase (N=102) | Anacetrapib 100 mg - Reversal Phase (N=196) | Placebo - Reversal Phase (N=95)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug resistance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anacetrapib 100 mg - Treatment Phase (N=203) | Placebo - Treatment Phase (N=102) | Anacetrapib 100 mg - Reversal Phase (N=196) | Placebo - Reversal Phase (N=95)
Diarrhoea (Gastrointestinal disorders) | 16 (19) | 9 (10) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 6 (7) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 20 (22) | 11 (11) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 40 (50) | 19 (21) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (26) | 4 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (19) | 6 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.